CLINICAL TRIAL: NCT04670302
Title: The Efficacy of Using Allogeneic Adipose-derived Mesenchymal Stem Cells and Human Amniotic Membrane (AAdMSC-HAM) Composite for Supraspinatus Tendon Repair Augmentation
Brief Title: Mesenchymal Stem Cells and Amniotic Membrane Composite for Supraspinatus Tendon Repair Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1208/KEPK/V/2019
Record Dates: First submitted 2020-12-08; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Supraspinatus Tear
Keywords: Supraspinatus rupture; Supraspinatus tear; Tendon repair; Tendon tissue engineering; Amniotic membrane; Mesenchymal stem cells

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Tendon repair) (Active Comparator): The control group will undergo tendon repair procedure only (without augmentation)
  Interventions: Procedure: Tendon repair procedure
- Experimental group (Tendon repair augmented with AAdMSC-HAM composite) (Experimental): The experimental group will undergo tendon repair procedure augmented with AAdMSC-HAM composite
  Interventions: Procedure: Tendon repair augmented with AAdMSC-HAM composite

INTERVENTIONS:
Procedure: Tendon repair procedure — Tendon repair procedure:
  1. Single senior surgeon (HS) will perform mini-open surgery to decompress the acromioplasty and repair the supraspinatus tendon.
  2. Splicing is achieved by installing screw-type anchors on the insertional footprint of the humeral head greater tuberosity.
  3. Then, double suturing of the supraspinatus tendon is performed.
  Arms: Control group (Tendon repair)
Procedure: Tendon repair augmented with AAdMSC-HAM composite — After double suturing of the supraspinatus tendon, the composite comprising freeze-dried HAM (2 cm x 2 cm x 0.002 cm) and AAdMSC (20 million cells) is placed on the upper surface of the splice and fixed with stitches at all four corners.
  Arms: Experimental group (Tendon repair augmented with AAdMSC-HAM composite)

SUMMARY:
This is a non-randomized clinical trial conducted in a single tertiary hospital which investigates the efficacy of allogeneic adipose-derived mesenchymal stem cells and human amniotic membrane (AAdMSC-HAM) composite for supraspinatus tendon repair augmentation

DETAILED DESCRIPTION:
Supraspinatus tendon tear is the most common factor causing shoulder pain, mainly resulting in discomfort and functional deficit in individuals over the age of 35. Supraspinatus tendon repair surgery represents one of the most widely performed types of orthopedic operation. Nevertheless, concerns persist regarding tendon-to-bone healing during the postoperative period. Despite advancements in surgical technique, re-tear of a previously repaired supraspinatus tendon is a fairly common complication, especially in a larger size tear. Such repair technique employing suture anchor devices alone has not yet produced functional results demonstrating both anatomical and biomechanical properties. Therefore, tendon tissue engineering using a combination of scaffolds, cells, and growth factors stimulation offers a potential solution as a biological augmentation in tendon repair.

Human amniotic membrane (HAM) has been widely used as a natural scaffold in tissue engineering due to many of its unique properties such as providing growth factors, cytokines and tissue inhibitors of metalloproteinases, adequate mechanical strength, and biocompatibility. Whereas, mesenchymal stem cells (MSCs) constitute one of the adult stem cells that promote replacement and repair of damaged tissue along with normal tissue turnover. These MSCs are seeded to the HAM scaffolds to biologically augment tendon repair, with MSCs acting as cytokines/growth factors to stimulate tissue repair. This approach serves as the foundation to conduct the present study. The investigators aim to investigate the efficacy of using allogeneic adipose-derived MSCs and human amniotic membrane (AAdMSC-HAM) composite for supraspinatus tendon repair augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from complete/total tear of supraspinatus tendon for a duration of fewer than 12 months
* Diagnosis is established based on clinical condition and ultrasonography or MRI examination

Exclusion Criteria:

* Patients with comorbid diseases: Diabetes Mellitus, Rheumatoid Arthritis, and other inflammatory diseases.
* Patients presenting with other related injuries, such as fractures or dislocation around the shoulder joint.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Active range of motion (AROM) pre-surgery | Pre-surgery
  Shoulder: flexion, extension, abduction, adduction, external rotation, internal rotation.
  The tests are performed by two blinded assessor, and expressed in degrees.
Active range of motion (AROM) at 12 months follow-up | 12 months
  Shoulder: flexion, extension, abduction, adduction, external rotation, internal rotation.
  The tests are performed by two blinded assessor, and expressed in degrees.

SECONDARY OUTCOMES:
Pain pre-surgery | Pre-surgery Outcome
  Measured by visual analogue scales (VAS). Patients are asked to described their level of pain from the scale 0 to 10 (0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, 7-9 indicating severe pain, and 10 indicating the worst, unbearable pain). The lower scores mean a better pain outcome
Pain at follow-up 12 months | 12 months
  Measured by visual analogue scales (VAS). Patients are asked to described their level of pain from the scale 0 to 10 (0 indicating no pain, 1-3 indicating mild pain, 4-6 indicating moderate pain, 7-9 indicating severe pain, and 10 indicating the worst, unbearable pain). The lower scores mean a better pain outcome
Disabilities of the Arm, Shoulder, and Hand (DASH) score pre-surgery | Pre-surgery
  DASH score is a self-assessment of symptoms and function of the entire upper extremity comprising 30 items. Each item consists of five levels of answers (1=no difficulty/symptoms, 2=mild difficulty/symptoms, 3=moderate difficulty/symptoms, 4=severe difficulty/symptoms, and 5=extreme difficulty (unable to do)/symptoms). The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability). Greater DASH scores reflect greater disability (worse outcome).
Disabilities of the Arm, Shoulder, and Hand (DASH) score at follow-up 12 months | 12 months
  DASH score is a self-assessment of symptoms and function of the entire upper extremity comprising 30 items. Each item consists of five levels of answers (1=no difficulty/symptoms, 2=mild difficulty/symptoms, 3=moderate difficulty/symptoms, 4=severe difficulty/symptoms, and 5=extreme difficulty (unable to do)/symptoms). The scores are then used to calculate a scale score ranging from 0 (no disability) to 100 (most severe disability). Greater DASH scores reflect greater disability (worse outcome).
Constant-Murley Score (CS) pre-surgery | Pre-surgery
  The scoring system records individual parameters and provides an overall clinical functional assessment. It consists of 4 domains: pain, activities of daily living (ADL), mobility, and power/strength. Pain and ADL are self-assessed, while all other items are assessed by the blinded examiner. A higher score shows a better function (100 as the best), while a lower score shows a worse function (0 as the worst).
Constant-Murley Score (CS) at follow-up 12 months | 12 months
  The scoring system records individual parameters and provides an overall clinical functional assessment. It consists of 4 domains: pain, activities of daily living (ADL), mobility, and power/strength. Pain and ADL are self-assessed, while all other items are assessed by the blinded examiner. A higher score shows a better function (100 as the best), while a lower score shows a worse function (0 as the worst).
Tear recurrence (re-tear) | Throughout the study duration (12 months), recorded as the first time complained by the patients (i.e. after "n" months).
  A systematic review (D'Ambrosi et al., 2019) showed that re-tear rates after rotator cuff repair with scaffolds were 17.97%. We hypothesize that the augmentation using HAM (as scaffold) seeded with AAdMSC would further lower the re-tear rates. We plan to record the recurrence of supraspinatus tendon tear (if any) based on radiographic evaluation with ultrasonography, which will then be confirmed with MRI. Ultrasonography provides an excellent anatomical evaluation of soft tissue which is able to assess any alterations during active locomotion. However, due to its user-dependent nature, we will also confirm the findings with MRI examination. Any grade of re-tear (grade I-III as evaluated by ultrasonography and confirmed with MRI) will be counted in and classified as "re-tear". When the patients do not complain about any symptoms of re-tear, we will record them as "no re-tear".

CONTACTS AND LOCATIONS:
Overall Officials: Heri Suroto, MD, PhD, Principal Investigator — Cell and Tissue Bank-Regenerative Medicine, Dr. Soetomo General Academic Hospital, Indonesia
Locations (1):
- Dr. Soetomo General Academic Hospital/ Department Orthopaedic & Traumatology Faculty of Medicine Universitas Airlangga, Surabaya, East Java, Indonesia